CLINICAL TRIAL: NCT03066934
Title: A Multicentered Study on Efficiency of Noninvasive Ventilation Procedures
Acronym: SAFE-NIV
Status: Completed | Type: Observational
Sponsor: Akdeniz University (Other)
Collaborators: Ankara University (Other); Cukurova University (Other); Dokuz Eylul University (Other); Ege University (Other); Izmir Katip Celebi University (Other); TC Erciyes University (Other); Marmara University (Other); Koç University (Other); Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Oguz Dursun, MD, Associate Professor, Akdeniz University
Other Study IDs: 70904504/525
Record Dates: First submitted 2017-02-03; First posted 2017-03-01 (Actual); Last update posted 2019-09-10 (Actual); Status verified 2019-09

CONDITIONS: Noninvasive Positive Pressure Ventilation; High Flow Nasal Cannula; Failure, Respiratory
Keywords: Noninvasive Positive Pressure Ventilation; Nasal high flow; Respiratory Failure; Childhood
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Days
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- NIV Failure Group: NIV Failure Group consisted of children who failed their noninvasive ventilation session and required intubation or re-intubation
  Interventions: Other: noninvasive ventilation respiratory support
- NIV success group: Children who successfully managed their noninvasive ventilation therapy
  Interventions: Other: noninvasive ventilation respiratory support

INTERVENTIONS:
Other: noninvasive ventilation respiratory support

SUMMARY:
Noninvasive ventilation (NIV) is an alternative form of ventilatory support in critical care encompassing different modes of ventilation such as continuous positive airway pressure (CPAP), bilevel positive airway pressure (BiPAP) and high flow nasal cannula ventilation. Although numerous studies on adults exit in literature, the aspects of this ventilatory support is limited in pediatric age groups. Early recognition of respiratory failure and initiation of NIV in a pediatric patient would positively affect prognosis by avoiding certain complications of endotracheal intubation and mechanical ventilation and adds certain advantages. Decreasing re-intubation rates for the ones who are extubated but necessitating further oxygen support is another advantage of NIV. Although numerous studies on adults exit in literature, the aspects of this ventilatory support is limited in pediatric age groups. Besides, success as well as failure and complication rates in pediatric age groups vary extensively. This multi-centered, prospective cohort study is planned to observe the epidemiologic perspectives of study group within underlying problems, success rates between different age groups, complication and re-intubation rates and finally its' effect on prognosis and long term survival in a year period. Hence we believe results of this study would allow us to improve our knowledge on using this technique, applying different modes and parameters appropriately and design criteria to guide clinician in deciding which group of patients would benefit from NIV techniques.

DETAILED DESCRIPTION:
Total of 9 pediatric critical care centers all across the country will collaborate at this study:

1. Akdeniz University Faculty of Medicine, Pediatric Critical Care Division
2. Cukurova University Faculty of Medicine, Pediatric Critical Care Division
3. Ege University Faculty of Medicine, Pediatric Critical Care Division
4. Ankara University Faculty of Medicine, Pediatric Critical Care Division
5. Ondokuz Mayis University Faculty of Medicine, Pediatric Critical Care Division
6. Erciyes University Faculty of Medicine, Pediatric Critical Care Division
7. Koc University Faculty of Medicine, Pediatric Critical Care Division
8. Dokuz Eylül University Faculty of Medicine, Pediatric Critical Care Division
9. Izmir Katip Celebi University Faculty of Medicine, Pediatric Critical Care Division Since nature of this study is an observational cohort, all noninvasively ventilated children from one month to eighteen years will be enrolled in this study. A three-page questionnaire is designed to collect data. The first page includes information on epidemiological data, underlying disease in terms of both acute and chronicle problems resulting in respiratory problems; the second page includes a multi-colon table to record vital signs (heart and respiratory rate, systemic and diastolic blood pressure), PRISM-III and Pediatric logistic organ dysfunction (PELOD) scores, Glasgow coma scale, blood gas values, ventilation parameters, necessity of sedation (if so, drugs used for sedation) and finally comfort pain scores. Data will be collected immediately prior to commencing NIV, the first, second and sixth hours; if NIV support continues over 24 hours, then daily data will be obtained up to five days. Last questionnaire page consists of data for clinical outcome, reason of NIV failure, necessity of re-intubation and if so timing of re-intubation.

Primary outcome of this study is to observe success rates in decreasing necessity of mechanical ventilation or re-intubation. Successfully managed children will also be evaluated for age groups, underlying disease as well as modes of delivery and ventilation parameters to define thresholds on decision of NIV success or failure. Secondary outcome is to evaluate the NIV failure in terms of pediatric age groups, underlying disease, rates of NIV-related complications. If a respiratory failure occurs, modes of delivery and ventilation parameters, usage of different masks, timing of failure decision according to patients' clinical data will be explored from collected data.

Each center will fill in the questionnaire according to patient data and every two months period data will be collected from collaborators. After one year period, statistical evaluation will be investigated by the principle investigators.

Below participants may observe the questionnaire form:

Form - I

1. Age (months):
2. Sex:
3. Weight (kg):
4. PRISM - III score
5. Which one of the following describes the underlying disease? i. What is the acutely-developed illness that required noninvasive ventilation? (Can be marked more than one option)

   1. Heart failure
   2. Pneumonia
   3. Bronchiolitis /Asthma
   4. Acute respiratory distress syndrome (ARDS)
   5. Sepsis
   6. Laryngeal stridor after extubation (or respiratory distress)
   7. Other (please describe) :

   ii. What is the chronic underlying disease (Primary disease which occurred previously) (can be marked more than one option)
   1. Neuromotor disease
   2. Metabolic disease
   3. Malignancy
   4. Congenital cardiac disease
   5. Chronic pulmonary disease
   6. Immune deficiency
   7. Other (please specify)
   8. No chronic underlying disease
6. What is the type of respiratory insufficiency?

   1. Hypoxemic (Type I)
   2. Hypercapnic (Type II)
7. Was the patient intubated before noninvasive ventilation?

   1. Yes
   2. No
8. If participant's answer is YES to previous question, please describe the length of intubation period (hours):
9. Which one of the following describes NIV device?

   1. Specific noninvasive ventilation device
   2. Conventional mechanical ventilator with the noninvasive mode
   3. High flow nasal cannula
   4. BIPAP device (without oxygen blender)
   5. Other:
10. Which one of the mask types did participant apply in the patient?

    1. Nasal mask
    2. Oronasal mask
    3. Full face mask
    4. Nasal prong (cannula)
    5. Endotracheal tube
    6. Other (please specify):

Form - II: Variables attached below will be recorded at initial, first, second, sixth, 24th, 48th, 72th, 96th, 120th hours.

* Respiratory rate
* Heart rate
* Systolic tension
* Mean tension
* Diastolic tension
* PRISM - III score
* PELOD score
* Glasgow coma score
* Blood gas (arterial/ venous/ capillary)
* Partial arterial oxygen concentration (PaO2) / Fraction of Inspired oxygen (FiO2)
* Oxygen saturation (SpO2) / Fraction of Inspired oxygen ( FiO2)
* Partial arterial carbon dioxide concentration (PaCO2)
* Power of Hydrogen (pH)
* Device Mode
* Inspiratory positive airway pressure (IPAP) value
* Expiratory positive airway pressure (EPAP) value
* Fraction of inspired oxygen (FiO2) value
* Inspiratory time (IT)
* Rise time value
* Tidal volume
* Leakage (%)
* Mandatory rate
* High flow rate
* Sedo-analgesia drugs and dosage
* Comfort score

Form - III

1. Please select your observation on NIV success.

   1. Patient had to be re-intubated after 48 hours of NIV.
   2. Patient was successfully withdrawn from NIV in 48 hours.
   3. Patient received noninvasive ventilation for ……………………days.
2. If participant's answer is 'A' to the previous question, please specify the reason of re-intubation below (can be marked more than once)

   1. Patient - ventilator asynchrony
   2. Face - mask mismatch
   3. Significant leakage percentage
   4. Progress to respiratory failure (can be marked more than once) (i) SpO2/FiO2<193 in 0-1 hour (ii) FiO2 necessity > %80 (iii) Blood gas power of hydrogen (pH) <7.25 in two hours (iv) Failure to achieve 10% expected decrease in respiratory rate at second and sixth hours (v) Increase in clinically observed respiratory effort (vi) Progression to severe ARDS (Oxygenation index > 8)
   5. Neurologically deteriorating patient (Glasgow coma score < 8 or deterioration over three units)
   6. Risk of aspiration or bulbar dysfunction (loss of swallowing)
   7. Hemodynamic instability
   8. Arrythmia
   9. Pneumothorax
   10. Other (please specify):
3. If participant observes a complication in the patient, please specify below (can be marked more than once).

   1. Loss of skin intact
   2. Pneumothorax
   3. Puking and aspiration pneumonia
   4. Hemodynamic instability
   5. Other (please specify): ……………….................
   6. No complication was observed.
4. Please specify the length of noninvasive ventilation ………………………….. (hours)
5. If patient received NIV breaks in a day, please write down the length of ventilation hours per day.

   Day 1:……………………………… Day 2: …………………………………...
6. What is clinical outcome of the patient after noninvasive ventilation support?

   1. Respiratory failure diminished and patient was discharged from Pediatric intensive care unit (PICU) after ……………. (days / hours) .
   2. Patient was discharged form PICU with home- style noninvasive device after …………… days/hours)
   3. Patient necessitated tracheostomy.
   4. Patient died of respiratory failure after ………………. days/hours.
7. What is the length of hospital discharge? (please specify): …………………….

ELIGIBILITY:
Inclusion criteria:

1. noninvasively ventilated children
2. age: 1 month - less than 18 years

Exclusion criteria: none

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: all noninvasively ventilated children from one month to eighteen years will be enrolled in this study
Sampling Method: Non-Probability Sample
Enrollment: 352 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
To determine the incidence of NIV failure in children requiring invasive mechanical ventilation | one year
  NIV failure is defined as necessity of endotracheal intubation due to respiratory insufficiency within 48 hours in children receiving noninvasive ventilation in pediatric critical care units. Statistical analysis will be performed according to answers to form-I question-6 and form-III question-1 in the questionnaire.
To determine the incidence of NIV failure as re-intubation within 48 hours. | 1 year
  NIV failure is also determined as re-intubation within 48 hours for those who were previously intubated and received noninvasive ventilation following extubation. Second primary outcome will be evaluated by Form - I question-6 and Form - III question-1.

SECONDARY OUTCOMES:
To determine the reasons resulting in NIV failure in children enrolled in the study | one year
  Reasons of NIV failure is classified as; patient - ventilator asynchrony, face-mask mismatch, significant leakage percentage, progression to respiratory insufficiency [SpO2/FiO2<193 within the first hour; FiO2 necessity > %80 within two hours; blood gas pH<7.25 within two hours; failure to achieve 10 % expected decrease in respiratory rate within sixth hours, increase in clinically observed respiratory effort or progression to severe ARDS (Oxygenation index > 8)], neurologically deteriorating patient (Glasgow coma score < 8 or a decrease in score more than three units), risk of aspiration or bulbar dysfunction (loss of swallowing), hemodynamic instability, presence of arrhythmia and pneumothorax. Underlying causes of NIV failure will be evaluated by answers to question-2 in Form III.
To explore complication rates directly related to noninvasive ventilation. | one year
  Complications related to noninvasive ventilation are loss of skin intact, development of pneumothorax, puking and related aspiration pneumonia, and hemodynamic instability. Form - III question 3 will enlighten the incidence and the variety of complications.
To observe NIV success for those who receive noninvasive ventilation over 48 hours | one year
  Evaluation of answers to Form III questions 4-5-6 will demonstrate the NIV success for those who receive noninvasive ventilation over 48 hours as the third secondary outcome. Daily ventilation breaks and length of noninvasive support per day (day 1 to day 5) will also be recorded by investigators to investigate the association of NIV success and noninvasive durations by applying multiple logistic regression analysis.
To explore prognosis of patients receiving noninvasive ventilation | one year
  Final secondary outcome will be the exploration of prognosis and the interactions between efficiency of noninvasive ventilation by length of intensive care unit and hospital stay and as well as mortality regarding answers to questions six and seven in Form -III.

CONTACTS AND LOCATIONS:
Overall Officials: Oguz Dursun, Asc. Prof., Study Director — Akdeniz University Faculty of Mediciane
Locations (2):
- Turkey (Türkiye) (2):
  - Akdeniz University Faculty of Medicine Department of Pediatrics Division of Pediatric Critical Care, Antalya
  - Akdeniz University Faculty of Medicine, Antalya

IPD SHARING:
Plan to Share IPD: No